CLINICAL TRIAL: NCT01940861
Title: Cerebral Oxymetry in Traumatic Brain Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Co-TBI; 2010/824 (Other Grant/Funding Number: OUS)
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Traumatic brain injury

SUMMARY:
Vasopressor for current treatment protocols for acute traumatic brain injury can lead to vasoconstriction and thus cerebral hypoperfusion that can be detected with cerebral oxymetry as a drop in SCO2.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute traumatic severe brain injury requiring neuro intensive care.
* The patient admitted must be at least 18 years of age and under 60 years.
* Intoxication is not an obstacle for inclusion as we believe this will not affect the recording in relation to our problem.

Exclusion Criteria:

* Traumatic injury in the frontal lobes corresponding to the area where ScO2 monitored.
* Patients in pharmacological studies.
* Patients with severe heart / lung / blood vessel diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: TBI
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Dosage of vasopressor | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway